CLINICAL TRIAL: NCT02950337
Title: Phase II Study of Stereotactic Body Radiation Therapy for Un-biopsied Early- Stage Non Small Cell Lung Cancer
Brief Title: Stereotactic Body Radiation Therapy for Un-biopsied Early- Stage Non Small Cell Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Matthew Harkenrider, Assistant Professor, Residency Program Director & Director of Brachytherapy, Loyola University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 208111; 208111102115 (Other: Loyola University IRB)
Record Dates: First submitted 2016-09-09; First posted 2016-11-01 (Estimated); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Unbiopsied Early Stage Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1: Peripherally Located Tumors (Experimental): Peripherally Located Tumors - SBRT
  Interventions: Radiation: Group 1: Peripherally Located Tumors
- Group 2: Peripherally Located Chest Wall Adjacent Tumors (Experimental): Peripherally Located Chest Wall Adjacent Tumors - SBRT
  Interventions: Radiation: Group 2: Peripherally Located Chest Wall Adjacent Tumors
- Group 3: Centrally Located Tumors (Experimental): Centrally Located Tumors - SBRT
  Interventions: Radiation: Group 3: Centrally Located Tumors

INTERVENTIONS:
Radiation: Group 1: Peripherally Located Tumors — Group 1: For peripherally located tumors patients will receive SBRT(Stereotactic Body Radiation Therapy) , 3 fractions of 18 Gy to a total dose of 54 Gy, with a minimum of 40 hours between each treatment fraction is required. ( Gy = Gray and is the unit used to measure the total amount of radiation a patient is exposed to)
  Arms: Group 1: Peripherally Located Tumors
Radiation: Group 2: Peripherally Located Chest Wall Adjacent Tumors — Group 2: For chest wall adjacent tumors patients will receive SBRT (Stereotactic Body Radiation Therapy) , 5 fractions of 12 Gy to a total dose of 60 Gy, with a minimum of 40 hours between each treatment fraction is required. ( Gy = Gray and is the unit used to measure the total amount of radiation a patient is exposed to)
  Arms: Group 2: Peripherally Located Chest Wall Adjacent Tumors
Radiation: Group 3: Centrally Located Tumors — Group 3: For central tumors patients will receive SBRT (Stereotactic Body Radiation Therapy) , 5 fractions of 10 Gy to a total dose of 50 Gy, with a minimum of 40 hours between each treatment fraction is required. ( Gy = Gray and is the unit used to measure the total amount of radiation a patient is exposed to)
  Arms: Group 3: Centrally Located Tumors

SUMMARY:
Lung cancer is the leading cause of cancer death in both men and women in the United States. In 2014, an estimated 224,210 men and women were diagnosed with carcinoma of the lung and bronchus, resulting in 159,260 deaths. Per the current National Comprehensive Cancer Network (NCCN) guidelines, the standard of care for early-stage non-small cell lung cancer (NSCLC) is lobectomy with lymph node dissection. Historically, medically inoperable early-stage NSCLC patients have been offered definitive external beam radiotherapy (EBRT) as primary management but, overall, studies have consistently shown poor patient outcomes. Stereotactic body radiation therapy (SBRT) is a technique which delivers very high doses of radiation per fraction over one to five fractions to precisely defined volumes with steep dose gradients. SBRT is commonly utilized for the treatment of biopsy-proven early stage NSCLC in the medically inoperable patient.

DETAILED DESCRIPTION:
This purpose of this study is to learn about the good and bad effects of treating early stage lung cancer without having a biopsy of the tumor. Participants in this research will receive a type of radiation treatment called Stereotactic Body Radiation Therapy (SBRT). This type of radiation is targeted directly at the tumor so that damage to surrounding normal tissue can be avoided. SBRT is often used in treating patients with biopsy proven early stage lung cancer who cannot have surgery for medical reasons. In this study, SBRT is considered experimental because the tumor has not been biopsied. SBRT for early-stage NSCLC has consistently proven to provide excellent local control and improved overall survival in the medically inoperable patient. The constancy of this finding over a variety of dose schedules confirms the robustness of SBRT. This study will utilize 54 Gy in 3 fractions delivered twice weekly for peripheral lesions. In order to respect the increased risk of adverse events our dose for centrally located lesions will be reduced to 50 Gy in 5 fractions delivered twice weekly and for chest wall or rib adjacent lesions will be 60 Gy in 5 fractions. These doses are consistent with Radiation Therapy Oncology Group (RTOG) 0236 for peripheral lesions and RTOG 0813 for central lesions and are both ≥100 Gy Biological Effective Dose (BED) as previously discussed . The investigators of this study routinely prescribe 60 Gy in 5 fractions for rib adjacent lesions.

The primary objective is to assess acute and chronic toxicities associated with SBRT of unbiopsied early-stage NSCLC.

Secondary objectives include:

To evaluate the disease specific outcomes of local control, lobar failure-free survival, regional/nodal failure-free survival, distant metastasis-free survival, disease-free survival, cause-specific survival, and overall survival associated with SBRT of unbiopsied early-stage NSCLC patients.

To evaluate Pulmonary Function Test (PFT) changes over time following SBRT of unbiopsied early-stage NSCLC patients.

To evaluate the patient's overall quality of life before and after treatment with SBRT of unbiopsied early-stage NSCLC patients.

ELIGIBILITY:
Inclusion Criteria

* • Presence of parenchymal lung nodule, without pathological diagnosis, highly suspicious for NSCLC as defined by at least one of the criteria below. Validated clinical prediction model estimates probability of malignancy is ≥ 85% or

  * Multidisciplinary tumor board determines patient's history, clinical findings, and radiographic findings are consistent with high probability of malignancy.

Medically-inoperable patient due to one of the criteria below

* Poor pulmonary function for resection including baseline Forced Expiratory Volume in 1 second (FEV1), FEV1 <50%, post-operative predicted FEV1<30% predicted, diffusion capacity <50%, baseline hypoxemia and/or hypercapnia. Patients with severe obstructive or restrictive lung disease will be eligible for inclusion.
* Pulmonary hypertension
* Cerebral, cardiac, or peripheral vascular disease
* Chronic heart disease
* Diabetes mellitus with end organ damage
* Age ≥75
* Patient declines surgery

Absence of pathological diagnosis due to one of the criteria below

* High risk of complications from transbronchial or transthoracic biopsy
* Biopsy was performed or attempted but with complications requiring abortion of procedure
* Biopsy was performed and non-diagnostic for malignancy but without other diagnosis to explain the clinical and radiographic findings
* Patient declines biopsy Stage T1-3, N0, M0 (AJCC Staging, 7th Ed.) based upon the following diagnostic workup
* History/Physical examination by an experienced thoracic cancer clinician (thoracic surgeon, interventional pulmonologist, medical oncologist, or radiation oncologist) within 4 weeks prior to registration
* Diagnostic imaging (CT and/or PET/CT) Serial computed tomography and/or positron emission tomography imaging clinically consistent with lung malignancy.
* CT scan with contrast (unless medically contraindicated) within 6 weeks of registration. The tumor dimensions will be measured on CT with greatest dimension ≤5cm.
* Whole body Positron Emission Tomography / Computerized Tomography (PET/CT) within 12 weeks of registration. Standard uptake value (SUV) must be available but no minimum SUV is required for inclusion.

No clinical or radiographic evidence of nodal disease or distant metastases No previous local therapy such as external beam radiotherapy, lobectomy, or sublobar resection.

Women of child-bearing potential must undergo pregnancy testing prior to enrollment on study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

* A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months.

Patients with prior history of malignancy are permitted registration but must not be undergoing active cytotoxic or biologically-targeted therapy, must be disease-free from any malignancy for the previous three years, and must not have any history of brain metastases with the following exceptions:

* Patients with history of basal cell carcinoma and/or squamous cell carcinoma may be permitted access within 3 years of being disease-free and is up to the discretion of the treating physicians
* Patients with any prior history of lung cancer may not participate in this study.

Age ≥ 18 years. Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* • Prior history of lung cancer.

  * Prior local therapy (surgery or radiotherapy) for the current, clinically-diagnosed NSCLC.
  * Patients receiving any other investigational agents.
  * Patients with a known history of malignancy with a disease-free interval <3 years prior to enrollment or a history of brain metastases
  * Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, severely symptomatic congestive heart failure, cardiac arrhythmia, or psychiatric illness/social situations that could limit compliance with study requirements.
  * Patients who are currently pregnant or nursing due to the potential for congenital abnormalities and potential harm to nursing infants.
  * Patients enrolled on a competing investigational study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Toxicity Evaluation | 104 weeks
  Radiation related acute and chronic pulmonary grade 3-5 toxicity as defined by Common Terminology Criteria for Adverse Events (CTCAE) v 4.0 Toxicity evaluations will be done at weekly on treatment visits and at follow up visits for up to 104 weeks.

SECONDARY OUTCOMES:
Disease Specific Outcomes | 104 weeks
  Patients will be classified at week 104 as having (1) disappearance of the treated lesion (i.e., complete response), (2) at least 30% decrease in the diameter of the treated lesion (i.e., partial response), (3) at least 20% increase in the diameter of the treated lesion (i.e., progressive disease), or (4) Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease (i.e., stable disease). Disease outcomes will be assessed during follow up exams up to 104 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Harkenrider, MD, Principal Investigator — Loyola University; Matthew Harkenrider, MD, Principal Investigator — Edward Hines Jr. VA Hospital
Locations (2):
- United States (2):
  - Edward Hines Jr, VA Hospital, Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Siegel R, Ma J, Zou Z, Jemal A. Cancer statistics, 2014. CA Cancer J Clin. 2014 Jan-Feb;64(1):9-29. doi: 10.3322/caac.21208. Epub 2014 Jan 7. PMID 24399786
- [Result] Qiao X, Tullgren O, Lax I, Sirzen F, Lewensohn R. The role of radiotherapy in treatment of stage I non-small cell lung cancer. Lung Cancer. 2003 Jul;41(1):1-11. doi: 10.1016/s0169-5002(03)00152-1. PMID 12826306
- [Result] Dosoretz DE, Katin MJ, Blitzer PH, Rubenstein JH, Salenius S, Rashid M, Dosani RA, Mestas G, Siegel AD, Chadha TT, et al. Radiation therapy in the management of medically inoperable carcinoma of the lung: results and implications for future treatment strategies. Int J Radiat Oncol Biol Phys. 1992;24(1):3-9. doi: 10.1016/0360-3016(92)91013-d. PMID 1324899
- [Result] Sibley GS, Jamieson TA, Marks LB, Anscher MS, Prosnitz LR. Radiotherapy alone for medically inoperable stage I non-small-cell lung cancer: the Duke experience. Int J Radiat Oncol Biol Phys. 1998 Jan 1;40(1):149-54. doi: 10.1016/s0360-3016(97)00589-0. PMID 9422571
- [Result] Zierhut D, Bettscheider C, Schubert K, van Kampen M, Wannenmacher M. Radiation therapy of stage I and II non-small cell lung cancer (NSCLC). Lung Cancer. 2001 Dec;34 Suppl 3:S39-43. doi: 10.1016/s0169-5002(01)00381-6. PMID 11740992
- [Result] Kupelian PA, Komaki R, Allen P. Prognostic factors in the treatment of node-negative nonsmall cell lung carcinoma with radiotherapy alone. Int J Radiat Oncol Biol Phys. 1996 Oct 1;36(3):607-13. doi: 10.1016/s0360-3016(96)00364-1. PMID 8948345
- [Result] Kaskowitz L, Graham MV, Emami B, Halverson KJ, Rush C. Radiation therapy alone for stage I non-small cell lung cancer. Int J Radiat Oncol Biol Phys. 1993 Oct 20;27(3):517-23. doi: 10.1016/0360-3016(93)90374-5. PMID 8226143
- [Result] Fakiris AJ, McGarry RC, Yiannoutsos CT, Papiez L, Williams M, Henderson MA, Timmerman R. Stereotactic body radiation therapy for early-stage non-small-cell lung carcinoma: four-year results of a prospective phase II study. Int J Radiat Oncol Biol Phys. 2009 Nov 1;75(3):677-82. doi: 10.1016/j.ijrobp.2008.11.042. Epub 2009 Feb 27. PMID 19251380
- [Result] Timmerman R, Paulus R, Galvin J, Michalski J, Straube W, Bradley J, Fakiris A, Bezjak A, Videtic G, Johnstone D, Fowler J, Gore E, Choy H. Stereotactic body radiation therapy for inoperable early stage lung cancer. JAMA. 2010 Mar 17;303(11):1070-6. doi: 10.1001/jama.2010.261. PMID 20233825
- [Result] Takeda A, Kunieda E, Sanuki N, Aoki Y, Oku Y, Handa H. Stereotactic body radiotherapy (SBRT) for solitary pulmonary nodules clinically diagnosed as lung cancer with no pathological confirmation: comparison with non-small-cell lung cancer. Lung Cancer. 2012 Jul;77(1):77-82. doi: 10.1016/j.lungcan.2012.01.006. Epub 2012 Jan 31. PMID 22300750
- [Result] Ricardi U, Filippi AR, Guarneri A, Giglioli FR, Ciammella P, Franco P, Mantovani C, Borasio P, Scagliotti GV, Ragona R. Stereotactic body radiation therapy for early stage non-small cell lung cancer: results of a prospective trial. Lung Cancer. 2010 Apr;68(1):72-7. doi: 10.1016/j.lungcan.2009.05.007. Epub 2009 Jun 24. PMID 19556022
- [Result] Gould MK, Maclean CC, Kuschner WG, Rydzak CE, Owens DK. Accuracy of positron emission tomography for diagnosis of pulmonary nodules and mass lesions: a meta-analysis. JAMA. 2001 Feb 21;285(7):914-24. doi: 10.1001/jama.285.7.914. PMID 11180735
- [Result] Gould MK, Donington J, Lynch WR, Mazzone PJ, Midthun DE, Naidich DP, Wiener RS. Evaluation of individuals with pulmonary nodules: when is it lung cancer? Diagnosis and management of lung cancer, 3rd ed: American College of Chest Physicians evidence-based clinical practice guidelines. Chest. 2013 May;143(5 Suppl):e93S-e120S. doi: 10.1378/chest.12-2351. PMID 23649456
- [Result] Herder GJ, van Tinteren H, Golding RP, Kostense PJ, Comans EF, Smit EF, Hoekstra OS. Clinical prediction model to characterize pulmonary nodules: validation and added value of 18F-fluorodeoxyglucose positron emission tomography. Chest. 2005 Oct;128(4):2490-6. doi: 10.1378/chest.128.4.2490. PMID 16236914
- [Result] Harkenrider MM, Bertke MH, Dunlap NE. Stereotactic body radiation therapy for unbiopsied early-stage lung cancer: a multi-institutional analysis. Am J Clin Oncol. 2014 Aug;37(4):337-42. doi: 10.1097/COC.0b013e318277d822. PMID 23660597
- [Result] Timmerman RD. An overview of hypofractionation and introduction to this issue of seminars in radiation oncology. Semin Radiat Oncol. 2008 Oct;18(4):215-22. doi: 10.1016/j.semradonc.2008.04.001. No abstract available. PMID 18725106
- [Result] Dunlap NE, Cai J, Biedermann GB, Yang W, Benedict SH, Sheng K, Schefter TE, Kavanagh BD, Larner JM. Chest wall volume receiving >30 Gy predicts risk of severe pain and/or rib fracture after lung stereotactic body radiotherapy. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3):796-801. doi: 10.1016/j.ijrobp.2009.02.027. Epub 2009 May 8. PMID 19427740